CLINICAL TRIAL: NCT06064981
Title: Behavioral Economic Approaches to Increase Naloxone Aquisition and Carrying in an Urban Environment
Brief Title: BE Intervention for Naloxone Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carolyn Cannuscio, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 831618
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Harm Reduction
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the control arm receive usual care. In this case they receive naloxone training only. The training involves a 1-hour in-person overdose recognition and reversal course, which addressed the following topics: the scope and nature of the opioid overdose epidemic nationally and locally in Philadelphia, signs of opioid overdose, strategies for approaching or interacting with a person who is suspected to have overdosed, administration of naloxone in its nasal spray formulation, what to expect after administering naloxone, legal considerations and Good Samaritan protection, and how and where to acquire naloxone.
- Text message nudges (Experimental): Participants in this arm receive text message nudges with salient messaging around overdose and naloxone. They also receive naloxone training.
  Interventions: Behavioral: Text message nudges
- Commitment contract (Experimental): Participants in this arm receive sign a commitment contract agreeing to obtain or carry naloxone. They also receive naloxone training.
  Interventions: Behavioral: Commitment contract

INTERVENTIONS:
Behavioral: Text message nudges — Fourteen text message "nudges," tailored to address specific barriers and concerns regarding naloxone acquisition and carrying. These barriers were identified using qualitative interviews conducted by the authors in prior studies. Examples included: optimism bias (e.g., beliefs that participants were unlikely to encounter someone who had overdosed in their daily lives), and identity bias (e.g., beliefs that participants were not the type of people who could save a life).
  Arms: Text message nudges
Behavioral: Commitment contract — In addition to the training, participants in the third arm were asked to sign commitment contracts, which had language in which they "committed" to carrying/acquiring naloxone.
  Arms: Commitment contract

SUMMARY:
The overall objective of this study is to use behavioral economics interventions to increase naloxone acquisition and carrying among participants who attend an opioid overdose reversal training.

DETAILED DESCRIPTION:
This study aims to use behavioral economics interventions to increase naloxone acquisition and carrying among participants who attend opioid overdose reversal training. The study consists of two distinct randomized controlled trials (Aim 2 and Aim 3) and has three primary objectives:

Aim 1: To diagnose behavioral bottlenecks to naloxone acquisition and carrying. This aim involves analyzing data from naloxone training sessions to identify barriers to acquiring and carrying naloxone. These barriers will be mapped to cognitive biases, such as optimism bias and overconfidence, and will inform the behavioral interventions in Aims 2 and 3.

Aim 2: To test the impact of a behavioral economics intervention on naloxone acquisition. This aim involves a randomized controlled trial with 60 participants. The intervention group will receive commitment pledges, acquisition plans, and tailored text message nudges to increase naloxone acquisition within one week of training. The control group will receive standard training. The primary endpoint is the time it takes for participants to acquire naloxone post-training.

Aim 3: To test the impact of a text nudge intervention on naloxone carrying. This aim also involves a randomized controlled trial, where all participants receive naloxone at the training. The intervention group will receive tailored text message nudges to encourage consistent naloxone carrying. The control group (n=30) will not receive these nudges. The primary endpoint is the consistency of naloxone carrying post-training.

ELIGIBILITY:
Inclusion Criteria:

* Living in the Philadelphia area
* Attended the study naloxone training.

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
Naloxone carrying | Proportion of successful naloxone check-ins at 14 random time points over a 4 week period post-intervention.
  Assessed by photo documentation via text message.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Cannuscio, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No